CLINICAL TRIAL: NCT01720641
Title: Partner Notification Strategies for STI Control in Urban Peru
Brief Title: Partner Notification Strategies for MSM in Peru
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Asociación Civil Impacta Salud y Educación, Peru (Other)
Responsible Party: Principal Investigator, Jesse Clark, Assistant Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K23MH084611 (NIH); IMP-478-2012 (Other: Instituto Nacional de Salud del Peru); K23MH084611 (NIH)
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Partner Notification Following STI Diagnosis
Keywords: MSM; Transgender Women; Partner Notification; Syphilis; Peru
MeSH Terms: conditions — Syphilis | interventions — Patient Portals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): Standardized partner notification counseling
- Internet Notification (Experimental): Standardized partner notification counseling and referral to internet-based partner referral website.
  Interventions: Behavioral: Internet
- Referral Card (Experimental): Standardized partner notification counseling and provision of 5 printed partner referral cards.
  Interventions: Behavioral: Referral Card
- Internet and Referral Card (Experimental): Standardized partner notification counseling and referral to internet-based partner referral website and provision of 5 printed partner referral cards.
  Interventions: Behavioral: Internet and Referral Card

INTERVENTIONS:
Behavioral: Internet — Referral and user instructions for Peru section of www.inspot.org partner notification website
  Arms: Internet Notification
Behavioral: Referral Card — 5 printed referral cards with information on syphilis signs, symptoms, diagnosis, treatment, and local resources.
  Arms: Referral Card
Behavioral: Internet and Referral Card — 5 printed referral cards with information on syphilis signs, symptoms, diagnosis, treatment, and local resources; Referral and user instructions for Peru section of www.inspot.org partner notification website.
  Arms: Internet and Referral Card

SUMMARY:
The goal of the proposed research is to assess new strategies for partner management and sexually transmitted infection (STI) control to reduce the spread of HIV-1 among men who have sex with men (MSM) in Latin America. The HIV epidemic in Peru remains concentrated within the core risk group of MSM. STI infection and re-infection are central to the continuation of the HIV epidemic among MSM in Peru. Development of improved strategies for partner notification and treatment will reduce the incidence and prevalence of STIs and ultimately reduce the incidence of HIV infection in this population. The first phase of this study used qualitative methods to explore attitudes and practices related to partner notification among MSM in Lima, Peru. Findings from the qualitative research were used to develop a quantitative survey instrument to assess partner notification decision-making processes and practices among MSM in Peru recently diagnosed with HIV or syphilis infection. Data from both quantitative and qualitative phases of the study have been used to develop a partner notification for MSM in Peru. Investigators plan to implement and assess the impact of the intervention on rates of partner notification following a diagnosis of syphilis among MSM in Lima, Peru. The investigators hypothesize that participants randomized to receive one or more partner notification tools will report a higher frequency of partner notification.

DETAILED DESCRIPTION:
Specific Aim: To assess the efficacy of internet- and referral card-based partner notification tools for the improvement of partner notification outcomes among MSM in Lima, Peru. As attitudes and behaviors related to partner notification vary within specific behavioral, social, and clinical contexts, interventions designed to improve partner notification outcomes must address the same contextual determinants to be effective. Partner notification tools based on electronic distribution of anonymous notification messages and/or patient-delivered referral cards are expected to increase notification rates in specific contexts.

Hypothesis: Provision of partner notification tools based on electronic and printed resources will improve reported and observed partner notification outcomes by overcoming barriers to notification including limited contact information, fear of disclosure, stigma, and lack of informational resources. Notification outcomes and use of notification tools will vary according to strategies of interpersonal communication reflected in the specific behavioral, social, and biomedical contexts of the individual, the partnership, and the STI diagnosed.

Participants will be selected for participation in the study depending on the findings of the EPT/Partner Notification Screening Protocol. Participants in the EPT/Partner Notification Screening Protocol diagnosed with new syphilis infection will be eligible for enrollment in the Partner Notification protocol.

I. Recruitment: Participants in the EPT/Partner Notification Screening Protocol who are diagnosed with syphilis based on physician interpretation of results of RPR assay and clinical history will be invited by the Study Counselor to participate in the Partner Notification Intervention Protocol.

II. Informed Consent: All potential subjects will receive an explanation of the study procedures and risks and benefits and asked to provide written Informed Consent. Participants will be given the opportunity to take the Informed Consent Document home for further review and decide at a later time if they wish to participate in the study.

III. Enrollment: Subjects who consent to participate in the Partner Notification Intervention Protocol will be randomized to either the experimental Partner Notification intervention or the Standard of Care (Partner Notification Counseling) arm.

IV Randomization: Eligible subjects who provide consent to participate will be randomly assigned to intervention or control groups using a random permuted block allocation (block size=7 in an alternating 4/3 ratio). Computer-generated randomization assignments will be stored in opaque, sealed envelopes opened at the time of allocation. Randomization assignments will be recorded and identified by the participant's numeric study code.

V. Intervention Delivery. Participants assigned to the experimental Partner Notification intervention will be provided with standard partner notification counseling as well as 5 printed referral cards with information about syphilis infection and a referral sheet for the Spanish language version of the inSPOT internet-based partner notification service (www.inspot.org). Referral cards will include printed material informing the recipient that they may have been exposed to syphilis, and will provide information on syphilis infection, including local resources for testing and treatment. The inSPOT website is a free internet-based notification service that offers anonymous automated e-mail partner notification services following an STI diagnosis. Users of the system select a diagnosis as well as a standardized notification message which they can personalized with their name and other messages if they desire. The user then enters the e-mail address(es) of the person(s) they wish to notify and the system delivers an automated e-mail notification to the person advising them of their potential exposure to an STI and advising them to seek STI testing. The notification also includes the address of the inSPOT website which contains additional information on HIV/STIs, risks for transmission, and resources for testing and treatment. Participants will be instructed on how to use both tools to assist them in the partner notification process.

Participants randomized to the control arm will receive standard partner notification counseling by study staff, without any supplemental notification tools.

Following delivery of the intervention, an appointment will be scheduled for participants to return to the research site in 1 month.

VI. Follow-up Evaluation. All participants will be asked to return to the study site 1 month after enrollment and randomization. At the Follow-up evaluation, participants will complete a brief survey (Partner Notification Follow-up Survey).

VII. Survey: Participants will complete a brief follow-up survey assessing their general partner notification behavior as well as the actual notification and treatment outcome for each of their three most recent partners, as well as factors that impeded and/or promoted partner notification and treatment. Participants will be asked to specify whether each partner was notified, whether they received antibiotic treatment and/or sought STI testing, the participant's degree of certainty of the outcomes, and the reasons why each partner was or was not notified and/or treated.

VIII. Confirmation of Partner Notification: In order to provide independent confirmation of participant-reported notification status, study staff will ask participants for permission to conduct third party partner notification and confirmation of reported notification status. Participants will be asked for permission to contact their recent partner(s) by telephone or e-mail to confirm the notification outcome. Subjects will be informed that they are not obligated to provide contact information for any of their partners. Subjects will also be informed that if they provide contact information for their partner(s), study staff will contact the person using the contact information provided and notify the person only that someone they recently had sex with has been diagnosed with syphilis, provide information on local sites offering free or low cost testing for HIV and STIs, and answer any questions the partner might have. Subjects will be informed that study staff will not reveal the participant's name or other identifying information to their partner(s). If the participant provides contact information for their partner(s), study staff will contact the person and provide third-party partner notification using an IRB-approved script. After completing the partner notification process, study staff will ask the partner only if they had previously been notified by a partner about an STI diagnosis ("Yes/No"). Partners will not be asked for any additional information.

IX. Qualitative Evaluation. A randomly selected subgroup of participants in the Partner Notification Intervention Protocol will be invited to participate in individual interviews about the partner notification process. Each participant will be asked to participate in two interviews, one following randomization and one following the Follow-up Visit. Participants will complete a separate informed consent process for the individual interview and will receive additional compensation for their participation.

X. Eligibility. A randomly selected subset of participants from the Partner Notification intervention protocol will be invited to participate in the individual qualitative interviews. Every fourth participant randomized will be invited to participate in an individual interview until reaching the projected qualitative study sample of 20 participants (10 each from the intervention and control arms). Participants will be asked to complete a separate informed consent document indicating their willingness to participate in a qualitative interview.

XI. Interview Conduct. Interviews will be conducted in Spanish in a private room by a trained interviewer. Interviews will be recorded and transcribed verbatim. Participants will be advised that they can stop the interview at any time and that they will be able to stop the tape and erase any response during the interview if they desire.

XII. Interview Content: Baseline interviews will focus on individual decision-making processes regarding partner notification in specific partnership contexts with a focus on the influence of: STI-related stigma and shame; the gender and sexual identity of participants and their partner(s); perceived power differentials within the partnership(s); patterns of communication within the partnership(s); and structural access to testing and treatment.

Follow-up interviews will discuss actual notification and treatment outcomes. Follow-up interviews will emphasize: barriers or catalysts to implementing notification decisions in specific partnership contexts; structural access to partner testing and treatment within local social, cultural, and economic contexts; and the effectiveness of the study's quantitative outcomes in accurately measuring participants' lived experiences.

Each interview is expected to last approximately 20-30 minutes. Audio recordings and transcripts of interviews will be identified by the participant's numeric study code and the date of the interview.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Male or biologically male at birth
3. Sexual contact (oral or anal intercourse) with a male or male-to-female transgender partner in the past 12 months
4. Diagnosis with syphilis infection

Exclusion Criteria:

1. Under 18 years of age
2. Unable to understand informed consent procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Self-Reported Partner Notification | 21 days
  Participant self-report of recent partner notification at 14-21 days of follow-up.

SECONDARY OUTCOMES:
Investigator-confirmed Partner Notification | 21 Days
  Participants who report notifying one or more of their three most recent partners will be asked for permission for the investigators to contact one or more of these partners to confirm notification outcomes. Partners who are successfully contacted and confirm prior partner notification will be defined as confirmed notifications.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse L Clark, MD, MSc, Principal Investigator — University of California, Los Angeles
Locations (1):
- Asociacion Civil Impacta Salud y Educacion, Lima, Peru

REFERENCES:
- [Derived] Clark JL, Segura ER, Oldenburg CE, Salvatierra HJ, Rios J, Perez-Brumer AG, Gonzales P, Sheoran B, Sanchez J, Lama JR. Traditional and Web-Based Technologies to Improve Partner Notification Following Syphilis Diagnosis Among Men Who Have Sex With Men in Lima, Peru: Pilot Randomized Controlled Trial. J Med Internet Res. 2018 Jul 3;20(7):e232. doi: 10.2196/jmir.9821. PMID 29970355
- [Derived] Braun HM, Segura ER, Lake JE, Gandhi M, Rios J, Villaran MV, Sanchez J, Lama JR, Clark JL. Individual and partnership factors associated with anticipated versus actual partner notification following STI diagnosis among men who have sex with men and/or with transgender women in Lima, Peru. Sex Transm Infect. 2018 Dec;94(8):607-610. doi: 10.1136/sextrans-2017-053292. Epub 2017 Nov 30. PMID 29191814